CLINICAL TRIAL: NCT05340400
Title: The Prevalence and Risk Factors of Irritable Bowel Syndrome Among Adults: A Multi-Centre Cross-sectional Study.
Brief Title: The Prevalence and Risk Factors of Irritable Bowel Syndrome Among Adults
Status: Completed | Type: Observational
Sponsor: University of Aleppo (Other)
Responsible Party: Principal Investigator, Ahmad Yamen Arnaout, Principal Investigator, University of Aleppo
Other Study IDs: PRIBS Study
Record Dates: First submitted 2022-04-15; First posted 2022-04-22 (Actual); Last update posted 2022-06-14 (Actual); Status verified 2022-06

CONDITIONS: Irritable Bowel Syndrome; Colonic Diseases, Functional
Keywords: Rome IV criteria; Colonic Diseases; Digestive System Diseases; Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome; Colonic Diseases, Functional; Colonic Diseases; Digestive System Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients diagnosed with IBS: Collaborators will use Rome IV criteria for diagnosing IBS, and then divide participants into those with and without the disease.
  Interventions: Other: ROME IV Criteria
- Patients not diagnosed with IBS: Collaborators will use Rome IV criteria for diagnosing IBS, and then divide participants into those with and without the disease.
  Interventions: Other: ROME IV Criteria

INTERVENTIONS:
Other: ROME IV Criteria — Collaborators will use Rome IV criteria for diagnosing IBS by the presence of the abdominal pain at least once a week in the last 3 months, in addition to at least two of the following: abdominal pain related to defecation, change in stool frequency, or shape.

SUMMARY:
This is a multicenter cross-sectional study on the prevalence of Irritable Bowel Syndrome and the risk factors associated with it. The Rome IV criteria is used for diagnosing IBS. A questionnaire-guided interview will be applied to all subjects.

DETAILED DESCRIPTION:
: Irritable Bowel Syndrome (IBS) is a common functional bowel disorder characterized by abdominal pain or discomfort associated with defecation or an altered bowel habit. IBS can be divided into four subtypes according to the predominant bowel pattern: diarrhea-predominant (IBS-D), constipation-predominant (IBS-C), and both diarrhea and constipation (IBS-M), and when a stool pattern cannot be categorized under any of the above three patterns (IBS-U).

For clinicians, diagnosis of IBS can be challenging because symptoms can be variable over time, and what makes it a real challenge is the absence of a gold diagnostic standard for this syndrome. That is why experts developed the Rome criteria in 2006, which is constantly revised. The latest update of these criteria was published in 2016 as Rome IV.

Unfortunately, studies have indicated higher rates of psychological comorbidity including suicidal ideation and depression among IBS patients, and a significant reduction in health-related quality of life, this negatively affects the productivity of the individual in society. Epidemiological studies of this syndrome have indicated a greater prevalence among women than men, and adolescents among other age groups.

However, despite these attempts by researchers to determine the prevalence patterns and risk factors for this syndrome, many of them are still not sufficiently defined. Hence, our study came to determine the prevalence and risk factors of Irritable Bowel Syndrome among adults.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer to participate in the study

Exclusion Criteria:

* Poorly-controlled hyperthyroidism
* Poorly-controlled hypothyroidism
* Poorly-controlled hyperparathyroidism
* Liver disease
* Paralysis
* Parasitic diseases (worms ...)
* Celiac disease
* Inflammatory bowel disease (Crohn's disease or Ulcerative colitis)
* Lactose intolerance
* Cancer or tumor in the digestive tract

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Community sample.
Sampling Method: Non-Probability Sample
Enrollment: 5500 (Actual)
Dates: Start 2022-04-25 (Actual); Primary Completion 2022-05-25 (Actual); Study Completion 2022-06-10 (Actual)

PRIMARY OUTCOMES:
The Prevalence of Irritable Bowel Syndrome | 30 days
  Collaborators will make an interview questions using ROME IV to diagnose IBS among adults.

SECONDARY OUTCOMES:
Physical activity as risk factor for IBS | 30 days
  Collaborators will use the World Health Organization questionnaire to classify the physical activity of the participants into good and poor physical activity.
Perceived Stress Scale as risk factor for IBS | 30 days
  It is the most widely used measure of global perceived stress, and a robust predictor of health and disease. The total score is calculated on the basis of the answers to a series of questions based on monthly stress, and the participant's health status. PSS is a summary measure of ten items (range 0-4 points for every item). It is classified into low (PSS 0-13), moderate (PSS 14-26), and high perceived stress (PSS 27-40).
Fatigue as risk factor for IBS | 30 days
  Fatigue will be measured using the Chalder Fatigue Scale (CFQ), a self-administered questionnaire for measuring the extent and severity of fatigue within both clinical and non-clinical, epidemiological populations. CFQ is a summary measure of eleven items (range 0-33)
Diet and weight questions as risk factor for IBS | 30 days
  Collaborators will use a questionnaire to determine the participant's predominant dietary pattern, feeding patterns and allergies
Habits as risk factor for IBS | 30 days
  Smoking, drinking alcohol, caffeine intake, and sleep pattern.

CONTACTS AND LOCATIONS:
Locations (2):
- Syria (2):
  - Ahmad Yamen Arnaout, Aleppo
  - University of Aleppo, Aleppo

IPD SHARING:
Plan to Share IPD: No
Not available to other researchers.

REFERENCES:
- [Background] Mearin F, Lacy BE, Chang L, Chey WD, Lembo AJ, Simren M, Spiller R. Bowel Disorders. Gastroenterology. 2016 Feb 18:S0016-5085(16)00222-5. doi: 10.1053/j.gastro.2016.02.031. Online ahead of print. PMID 27144627
- [Background] Longstreth GF, Thompson WG, Chey WD, Houghton LA, Mearin F, Spiller RC. Functional bowel disorders. Gastroenterology. 2006 Apr;130(5):1480-91. doi: 10.1053/j.gastro.2005.11.061. PMID 16678561
- [Background] Drossman DA, Morris CB, Hu Y, Toner BB, Diamant N, Leserman J, Shetzline M, Dalton C, Bangdiwala SI. A prospective assessment of bowel habit in irritable bowel syndrome in women: defining an alternator. Gastroenterology. 2005 Mar;128(3):580-9. doi: 10.1053/j.gastro.2004.12.006. PMID 15765393
- [Background] Palsson OS, Baggish JS, Turner MJ, Whitehead WE. IBS patients show frequent fluctuations between loose/watery and hard/lumpy stools: implications for treatment. Am J Gastroenterol. 2012 Feb;107(2):286-95. doi: 10.1038/ajg.2011.358. Epub 2011 Nov 8. PMID 22068664
- [Background] Zamani M, Alizadeh-Tabari S, Zamani V. Systematic review with meta-analysis: the prevalence of anxiety and depression in patients with irritable bowel syndrome. Aliment Pharmacol Ther. 2019 Jul;50(2):132-143. doi: 10.1111/apt.15325. Epub 2019 Jun 3. PMID 31157418
- [Background] Gralnek IM, Hays RD, Kilbourne A, Naliboff B, Mayer EA. The impact of irritable bowel syndrome on health-related quality of life. Gastroenterology. 2000 Sep;119(3):654-60. doi: 10.1053/gast.2000.16484. PMID 10982758
- [Derived] Arnaout AY, Nerabani Y, Douba Z, Kassem LH, Arnaout K, Shabouk MB, Zayat H, Mayo W, Bezo Y, Arnaout I, Yousef A, Zeina MB, Aljarad Z; PRIBS Study Team. The prevalence and risk factors of irritable bowel syndrome (PRIBS study) among adults in low- and middle-income countries: A multicenter cross-sectional study. Health Sci Rep. 2023 Oct 4;6(10):e1592. doi: 10.1002/hsr2.1592. eCollection 2023 Oct. PMID 37808932